CLINICAL TRIAL: NCT06654167
Title: Acute Effects of Cold Exposure on Cognitive Function and Underlying Mechanism
Brief Title: Acute Effects of Cold Exposure on Cognitive Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Renjie Chen, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB#2024-10-1168
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Function
Keywords: Low temperature; Randomized controlled trial; Cognitive function
MeSH Terms: interventions — Cold Temperature; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low temperature (15℃) group (Experimental): Subjects in the exposure group will be exposed to low temperature (15℃) for about 2 hours in a chamber.
  Interventions: Other: Low temperature (15℃) group
- Moderate temperature (22℃) group (Experimental): Subjects in the exposure group will be exposed to moderate temperature (22℃) for about 2 hours in a chamber.
  Interventions: Other: Moderate temperature (22℃) group

INTERVENTIONS:
Other: Low temperature (15℃) group — The exposure group will be exposed to low temperature (15℃) in a chamber for about 2 hours, resting during the whole period.
  Arms: Low temperature (15℃) group
Other: Moderate temperature (22℃) group — The exposure group will be exposed to thermoneutral temperature (22℃) in a chamber for about 2 hours, resting during the whole period.
  Arms: Moderate temperature (22℃) group

SUMMARY:
This is a randomized controlled human exposure crossover study. Investigators aims to assess the acute effects of low-temperature exposure on cognitive function and the underlying mechanisms.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled human exposure crossover study among about 40 healthy young adults in Shanghai, China. Each subject will be exposed twice: once to the low temperature (15℃) and once to the moderate temperature (22℃) in a chamber for about 2 hours. During the exposure session, each subject will be requested to rest. Health examinations will be conducted immediately prior to exposure, during the period of exposure, and after exposure. Health examinations include cognitive function tests and magnetic resonance imaging. Investigators plan to collect blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during the study period;
* Body mass index > 18.5 and ≤ 28;
* right-handed;
* receiving or having received higher education;
* with the ability to read and understand Chinese smoothly.

Exclusion Criteria:

* Smoking and alcohol abuse;
* Current drug and dietary supplements intake;
* Subjects with allergic diseases, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular diseases, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory diseases, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic diseases, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects who have a history of major surgery due to the cardiovascular, cerebrovascular, respiratory, or neurological diseases;
* Subjects with neurologic disorders, such as stroke, traumatic brain injury, epilepsy, and schizophrenia;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Subjects with color vision disabilities.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Results of Stroop Tests | before exposure and immediately after the exposure session
  Investigators plan to measure the changes of cognitive function using Stroop Test. The time taken to complete the test could reflect cognitive function, and a shorter time means better cognitive function.

SECONDARY OUTCOMES:
Results of simple reaction time | before exposure and immediately after the exposure session
  Investigators plan to measure the changes of cognitive function using visual memory test
Activated brain regions demonstrating neural activity related to the high temperature exposure | 1 hour after exposure session
  Investigators plan to measure brain activity associated with high temperature exposure by magnetic resonance imaging (MRI). Brain imaging data will be extracted from MRI data. The fractional amplitude of low frequency fluctuation (fALFF) would be extracted to reflect neural activity of brain regions.
Activated brain regions demonstrating neural connectivity related to the high temperature exposure | 1 hour after exposure session
  Investigators plan to measure brain activity associated with high temperature exposure by magnetic resonance imaging (MRI). Brain imaging data will be extracted from MRI data. The degree of centrality (DC) would be extracted to reflect neural connectivity of brain regions.
Activated brain regions demonstrating neural synchronization related to the high temperature exposure | 1 hour after exposure session
  Investigators plan to measure brain activity associated with high temperature exposure by magnetic resonance imaging (MRI). Brain imaging data will be extracted from MRI data. The regional homogeneity (ReHo) would be extracted to reflect neural synchronization of brain regions.
Changes of skin temperature | Skin temperature will be examined during the 2-hour exposure session (i.e., 1:00 P.M. to 3:00 P.M. on the day of the exposure session)
  The changes of wrist skin temperature will be measured

OTHER OUTCOMES:
Differences in RNA expression levels detected in serum transcriptomics between the two exposures | 1 hour after the exposure session
  Illumina-based transcriptomics is non-targeted. The study is to find the differentially expressed exosome RNA in serum after low temperature exposure
Change in brain-derived neurotrophic factor (BDNF) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of BDNF in blood.
Change in glial cell line-derived neurotrophic factor (GDNF) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of GDNF in blood.
Change in γ-aminobutyric acid (GABA) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of GABA in blood.
Change in Interleukin-1β (IL-1β) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of IL-1β in blood.
Change in Interferon-β (IFN-β) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of IFN-β in blood.
Change in glutathione (GSH) concentrations | 1:00 P.M. on the day of the exposure session, 1 hour after the exposure session
  Change in the concentrations of GSH in blood.
Changes of the scores of thermal sensation questionnaires | before exposure and immediately after the exposure session
  Changes of scores of thermal sensation questionnaires which ranged from -5 to 5. Zero score refers to the thermal comfort sensation. Higher scores refer to more uncomfortable sensations of hot. Lower scores refer to more uncomfortable sensations of cold.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Study Director — Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT06654167/SAP_000.pdf